CLINICAL TRIAL: NCT00842608
Title: Pharmacological Management of Delirium
Acronym: PMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, MALAZ BOUSTANI, Principal Investigator, Regenstrief Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0145; R01AG034205 (NIH)
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Delirium; Cognitive Impairment
Keywords: confusion; dementia
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Confusion; Dementia | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Haloperidol Eligible Intervention (Experimental): 0.5-1mg Haloperidol Q8h for 7 days, reduced exposure to anticholinergics, reduced exposure to benzodiazepines
  Interventions: Behavioral: Reduced exposure to anticholinergics; Procedure: Reduced exposure to benzodiazepines; Drug: Haloperidol
- Haloperidol Eligible Usual Care (Active Comparator): Usual care
  Interventions: Procedure: Usual care
- Haldol-Ineligible Arm (Experimental): Haldol-Ineligible arm for patients with contraindications for Haldol, unresolvable prolonged QTc, history of torsades de pointes, or history of seizures.
  Patients are randomized and will still receive:
  reduced exposure to anticholinergics, reduced exposure to benzodiazepines
  Interventions: Behavioral: Reduced exposure to anticholinergics; Procedure: Reduced exposure to benzodiazepines
- Haldol Ineligible Usual Care (Active Comparator): Usual Care
  Interventions: Procedure: Usual care

INTERVENTIONS:
Behavioral: Reduced exposure to anticholinergics — Using the computerized support, physicians will be notified if they attempt to prescribe a patient a medication with anticholinergic properties and will be given a safe alternative to the drug.
  Patients who are in the non-haldol arm will have their medical records manually reviewed by the study pharmacist as the computerized support is not set to differentiate between patients who can & cannot receive Haldol
  Arms: Haldol-Ineligible Arm; Haloperidol Eligible Intervention
Procedure: Reduced exposure to benzodiazepines — Tapering exposure to benzodiazepines by 50% over the first 48 hours after mechanical ventilation, complete stop by discharge; no benzodiazepine orders for patients not requiring mechanical ventilation
  Arms: Haldol-Ineligible Arm; Haloperidol Eligible Intervention
Drug: Haloperidol — 0.5 to 1 mg haloperidol every 8 hours via oral or parenteral route for a total of seven days or until discharge from the hospital
  Other Names: Haldol
  Arms: Haloperidol Eligible Intervention
Procedure: Usual care — May include use of typical and atypical neuroleptics, benzodiazepines, and other sedatives to manage the symptoms of delirium
  Arms: Haldol Ineligible Usual Care; Haloperidol Eligible Usual Care

SUMMARY:
The purpose of this study is to develop and test the feasibility of using a specific pharmacological protocol to reduce delirium burden among older adults in the Intensive Care Unit (ICU). The study will test the efficacy of a pharmacological intervention in reducing delirium severity and duration as well as length of stay and mortality compared to usual care.

DETAILED DESCRIPTION:
In 2005, approximately 2.7 million Americans aged 65 and older spent at least one day in the intensive care unit (ICU), costing Medicare an estimated $27.5 billion. It is estimated that while hospitalized, up to 80% of these older ICU patients had delirium, an acute brain failure that is an independent predictor of morbidity and mortality which often goes unrecognized. Older adults with delirium are more prone to falls, injuries, pressure ulcers and restraints, complications which may also contribute to prolonged ICU and hospital length of stay, higher mortality rates, poorer functional status, limited rehabilitation, increased institutionalization, and higher health care costs. The literature supports treatment with a combination of a reduction in the use of benzodiazepines and anticholinergics and the use of low-dose neuroleptics such as haloperidol. However, there have been no randomized controlled trials evaluating the efficacy of this approach on reducing delirium severity, duration, and complications.

Building upon the e-CHAMP study, ("Enhancing Care for Hospitalized Older Adults With Memory Problems;" see NCT00182832), a recently completed quality improvement project tested the effectiveness of cognitive screening coupled with computerized decision support in reducing delirium and other hospital-related complications among 424 older adults hospitalized on the medical wards, which found that many of the older adults entering the study had already experienced delirium in the ICU prior to their transfer to the wards. This study will test a pharmacologic intervention that allows a more targeted approach to the care of older adults with delirium while still recognizing the clinicians' role in controlling symptoms and providing intensive care.

The hypothesis is that patients in the intervention arm as compared to usual care will have:

* reduced delirium severity, as measured by the Delirium Rating Scale (DRS-R-98), at one week following randomization or hospital discharge
* fewer hospital days with delirium or coma as determined by the Confusion Assessment Method in the ICU (CAM-ICU)
* shorter hospital lengths of stay
* lower ICU, hospital, and 30-day mortality

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Hospitalized on an ICU ward
* Delirium based on the RASS and the CAM-ICU assessments at any day during ICU stay
* English speaking

Exclusion Criteria:

* Admitted directly to a regular non-ICU ward
* Previously enrolled in the study
* Not eligible for delirium assessment as determined by RASS scores
* Prior history of severe mental illness
* Alcohol-related delirium
* Pregnant or nursing
* Have had an aphasic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2009-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malaz Boustani, MD, Principal Investigator — Indiana University School of Medicine
Locations (3):
- United States (3):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana
  - University Hospital, Indianapolis, Indiana

REFERENCES:
- [Derived] Wang S, Perkins AJ, Chi R, Yates BA, Khan SH, Gao S, Boustani M, Khan BA. Risk factors for dementia in older intensive care unit (ICU) survivors. Alzheimers Dement. 2024 Jan;20(1):278-287. doi: 10.1002/alz.13423. Epub 2023 Aug 17. PMID 37589315
- [Derived] Ortiz D, Lindroth HL, Braly T, Perkins AJ, Mohanty S, Meagher AD, Khan SH, Boustani MA, Khan BA. Delirium severity does not differ between medical and surgical intensive care units after adjusting for medication use. Sci Rep. 2022 Aug 24;12(1):14447. doi: 10.1038/s41598-022-18429-9. PMID 36002562
- [Derived] Lindroth H, Khan BA, Carpenter JS, Gao S, Perkins AJ, Khan SH, Wang S, Jones RN, Boustani MA. Delirium Severity Trajectories and Outcomes in ICU Patients. Defining a Dynamic Symptom Phenotype. Ann Am Thorac Soc. 2020 Sep;17(9):1094-1103. doi: 10.1513/AnnalsATS.201910-764OC. PMID 32383964
- [Derived] Khan BA, Perkins AJ, Campbell NL, Gao S, Farber MO, Wang S, Khan SH, Zarzaur BL, Boustani MA. Pharmacological Management of Delirium in the Intensive Care Unit: A Randomized Pragmatic Clinical Trial. J Am Geriatr Soc. 2019 May;67(5):1057-1065. doi: 10.1111/jgs.15781. Epub 2019 Jan 25. PMID 30681720
- [Derived] Campbell NL, Khan BA, Farber M, Campbell T, Perkins AJ, Hui SL, Abernathy G, Buckley J, Sing R, Tricker J, Zawahiri M, Boustani MA. Improving delirium care in the intensive care unit: the design of a pragmatic study. Trials. 2011 Jun 6;12:139. doi: 10.1186/1745-6215-12-139. PMID 21645330

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 551 patients were consented into the study. After completing the consent and randomization, 6 patients withdrew from the study and were included in intention-to-treat analysis. 545 patients completed the protocol.
Groups:
- Haloperidol Eligible Intervention: 0.5-1mg Haloperidol Q8h for 7 days, reduced exposure to anticholinergics, reduced exposure to benzodiazepines
  Reduced exposure to anticholinergics: Using the computerized support, physicians will be notified if they attempt to prescribe a patient a medication with anticholinergic properties and will be given a safe alternative to the drug.
  Patients who are in the non-haldol arm will have their medical records manually reviewed by the study pharmacist as the computerized support is not set to differentiate between patients who can & cannot receive Haldol
  Reduced exposure to benzodiazepines: Tapering exposure to benzodiazepines by 50% over the first 48 hours after mechanical ventilation, complete stop by discharge; no benzodiazepine orders for patients not requiring mechanical ventilation
  Haloperidol: 0.5 to 1 mg haloperidol every 8 hours via oral or parenteral route for a total of seven days or until discharge from the hospital
- Haldol-Ineligible Arm: Haldol-Ineligible arm for patients with contraindications for Haldol, unresolvable prolonged QTc, history of torsades de pointes, or history of seizures.
  Patients are randomized and will still receive:
  reduced exposure to anticholinergics, reduced exposure to benzodiazepines
  Reduced exposure to anticholinergics: Using the computerized support, physicians will be notified if they attempt to prescribe a patient a medication with anticholinergic properties and will be given a safe alternative to the drug.
  Patients who are in the non-haldol arm will have their medical records manually reviewed by the study pharmacist as the computerized support is not set to differentiate between patients who can & cannot receive Haldol
  Reduced exposure to benzodiazepines: Tapering exposure to benzodiazepines by 50% over the first 48 hours after mechanical ventilation, complete stop by discharge; no benzodiazepine orders for patients not requiring mechanical ventilation
Period: Overall Study
Arm/Group | Haloperidol Eligible Intervention | Haloperidol Eligible Usual Care | Haldol-Ineligible Arm | Haldol Ineligible Usual Care
Started | 174 | 177 | 99 | 101
Completed | 170 | 176 | 99 | 100
Not Completed | 4 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol Eligible Intervention | Haloperidol Eligible Usual Care | Haldol-Ineligible Arm | Haldol Ineligible Usual Care | Total
Number analyzed (Participants) | 174 | 177 | 99 | 101 | 551
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 112 | 114 | 57 | 59 | 342
  >=65 years | 62 | 63 | 42 | 42 | 209
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 86 | 65 | 53 | 302
  Male | 76 | 91 | 34 | 48 | 249
Region of Enrollment [Number; unit: participants]
  United States | 174 | 177 | 99 | 101 | 551

OUTCOME MEASURES:

1. Primary Outcome: Days Free of Delirium and Coma
Time Frame: Admission through day 8 of stay
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Haloperidol Eligible Intervention | Haloperidol Eligible Usual Care | Haldol-Ineligible Arm | Haldol Ineligible Usual Care
Number analyzed (Participants) | 174 | 177 | 99 | 101
days | 4 [2 to 7] | 5 [1 to 7] | 4 [1 to 7] | 5 [2 to 7]

2. Secondary Outcome: Hospital Length of Stay Post Randomization
Time Frame: Participants were followed for the duration of hospital stay, an average of 11 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Haloperidol Eligible Intervention | Haloperidol Eligible Usual Care | Haldol-Ineligible Arm | Haldol Ineligible Usual Care
Number analyzed (Participants) | 174 | 177 | 99 | 101
days | 20.2 (33.5) | 18.6 (31.6) | 18.8 (17.1) | 14.9 (11.8)

3. Secondary Outcome: Mortality
Time Frame: ICU, in-hospital, 30-days post hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol Eligible Intervention | Haloperidol Eligible Usual Care | Haldol-Ineligible Arm | Haldol Ineligible Usual Care
Number analyzed (Participants) | 174 | 177 | 99 | 101
Participants | 20 | 32 | 11 | 8

ADVERSE EVENTS:
Arm/Group | Haloperidol Eligible Intervention | Haloperidol Eligible Usual Care | Haldol-Ineligible Arm | Haldol Ineligible Usual Care
Serious Adverse Events (participants affected / at risk) | 45/174 | 57/177 | 27/99 | 22/101
Other Adverse Events (participants affected / at risk) | 87/174 | 82/177 | 63/99 | 59/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Haloperidol Eligible Intervention (N=174) | Haloperidol Eligible Usual Care (N=177) | Haldol-Ineligible Arm (N=99) | Haldol Ineligible Usual Care (N=101)
Patients with CNS (Nervous system disorders) | 5 | 7 | 4 | 2
Patients with Cardiovascular (Cardiac disorders) | 14 | 20 | 10 | 9
Patients with Respiratory (Respiratory, thoracic and mediastinal disorders) | 23 | 31 | 11 | 12
Patients with GI (Gastrointestinal disorders) | 6 | 6 | 3 | 3
Patients with GU (Renal and urinary disorders) | 7 | 4 | 0 | 4
Patients with Skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0
Patients with Hepatic (Hepatobiliary disorders) | 4 | 3 | 0 | 0
Patients with Hematologic (Blood and lymphatic system disorders) | 12 | 14 | 3 | 3
Patients with Endocrine (Endocrine disorders) | 1 | 1 | 0 | 0
Patients with Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Other (Investigations) | 7 | 0 | 4 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Haloperidol Eligible Intervention (N=174) | Haloperidol Eligible Usual Care (N=177) | Haldol-Ineligible Arm (N=99) | Haldol Ineligible Usual Care (N=101)
General Events (General disorders) | 87 | 82 | 63 | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No